CLINICAL TRIAL: NCT02513719
Title: XIENCE PRIME SV Everolimus Eluting Coronary Stent Japan Post Marketing Surveillance
Brief Title: XIENCE PRIME SV Everolimus Eluting Coronary Stent Japan Post Marketing Surveillance (XIENCE PRIME SV Japan PMS)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-303
Record Dates: First submitted 2015-07-17; First posted 2015-08-03 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2021-04

CONDITIONS: Ischemic Heart Disease; Angina Pectoris; Coronary Artery Disease; Coronary Artery Occlusion; Myocardial Ischemia
Keywords: drug eluting stent; stent; real world
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Coronary Artery Disease; Coronary Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- XIENCE PRIME SV Everolimus Eluting Coronary Stent: Patients receiving XIENCE PRIME SV Everolimus Eluting Coronary Stent
  Interventions: Device: XIENCE PRIME SV Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE PRIME SV Everolimus Eluting Coronary Stent — Patients receiving XIENCE PRIME SV Everolimus Eluting Stent

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of XIENCE PRIME SV in real world practice in Japanese hospitals.

DETAILED DESCRIPTION:
Based on Good Post-marketing Study Practice (GPSP) regulation, general patient population with ischemic heart disease who are eligible for treatment with XIENCE PRIME SV Everolimus Eluting Stent will be registered, with no particular inclusion/exclusion criteria, and may be eligible for angiographic follow-up at eight months and clinical follow-up at one year.

ELIGIBILITY:
* Patient informed consent is required for registration of this PMS. In cases where patient informed consent (or providing some type of information) is required for PMS per the participating site policy, the Sponsor will cooperate as needed.
* If it is known at the time of index procedure that the patient is not able to return for the 8-month follow-up visit for angiogram and for the 1-year clinical follow-up, then the patient should not be registered in the PMS.
* Patients who are treated (stent delivery system inserted into the body) by XIENCE PRIME SV will be registered (including provisional stenting for side branch treatment but excluding bail-out only use).

  * The observations will be compiled on a per-patient basis even if multiple stents are implanted during the index procedure.
  * A patient whose side-branch is treated by XIENCE PRIME SV can be registered. In such a case, main vessel should be treated by XIENCE PRIME.
  * A patient who are treated by other drug eluting stent (DES) for planned stent and XIENCE PRIME SV for bail-out purpose cannot be registered.
  * Additional revascularization procedures as a part of adverse event treatment and planned staged procedures will not be considered as another registration, or adverse events.
  * A patient who is treated, but failed to be implanted by XIENCE PRIME SV and finally treated by other devices only (No XIENCE PRIME SV are implanted) must also be registered. In such a case, only the stent information, device deficiency information and reportable adverse events related to the PRIME stent, if any, are required to be captured. Follow-up of the patient who does not receive any XIENCE PRIME SV stent is not required.
* A patient may have another lesion(s) that may be treated by larger diameter stent(s). In such a case, treatment by XIENCE PRIME is preferable. Lesion(s) treated by other than XIENCE PRIME is not considered as the target lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General patient population with ischemic heart disease in Japan who are eligible for treatment with XIENCE PRIME SV Everolimus Eluting Stent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kozuma, MD, Study Chair — Teikyo University Hospital, Tokyo
Locations (33):
- Japan (33):
  - Kimitsu Chuo Hospital, Chiba
  - Kokura Memorial Hospital, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka
  - Hoshi general hospital, Fukushima
  - Tsuchiya General Hospital, Hiroshima
  - Hyogo Prefectural Amagasaki Hospital, Hyōgo
  - Tsukuba Medical Center Hospital, Ibaraki
  - Ishikawa Prefectual Central Hospital, Ishikawa
  - Shonan Kamakura General Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto Chuo Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Miyazaki City-Gun Ishikai Hospital, Miyazaki
  - Kansai Rosai Hospital, Nagoya
  - Nagoya Daini Red Cross Hospital, Nagoya
  - Heart disease center Sakakibara hospital, Okayama
  - Kurashiki Central Hospital, Okayama
  - Sakurabashi Watanabe Hospital, Osaka
  - Osaka police hospital, Osaka
  - Osaka University Hospital, Osaka
  - Tokorozawa Heart Center, Saitama
  - Tokeidai memorial hospital, Sapporo
  - JCHO Hokkaido Hospital, Sapporo
  - Hokkaido Ohno hospital, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Okamura memorial hospital, Shizuoka
  - Tokushima Red Cross Hospital, Tokushima
  - Mitsui Memorial Hospital, Tokyo
  - Toranomon hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Teikyo University Hospoital, Tokyo
  - Showa University Fujigaoka hospital, Yokohama
  - Saiseikai Yokohama City Tobu Hospital, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 312 subjects were enrolled from 30 sites. The enrollment period was from May 13, 2013 to March 25, 2014.
Period: At 8 Months Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 312
Completed | 312
Not Completed | 0
Period: At 1 Year Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 312
Completed | 305
Not Completed | 7
Period: At 2 Years Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 305
Completed | 300
Not Completed | 5
Period: At 3 Years Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 300
Completed | 289
Not Completed | 11
Period: At 4 Years Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 289
Completed | 273
Not Completed | 16
Period: At 5 Years Clinical Follow-up
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Started | 273
Completed | 254
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: 312 patients from 30 sites were treated with PRIME SV
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 235
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 312

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stent Thrombosis: Acute
Description: Stent/Scaffold Thrombosis (per ARC): Stent/Scaffold Thrombosis should be reported as a cumulative value over time and at various individual time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timing:
  Acute stent thrombosis: 0 to 24 hours after stent implantation
Time Frame: 0-24 hours post stent implantation
Population: Intent-To-Treat Population set (ITT). The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 1

2. Primary Outcome: Number of Participants With Stent Thrombosis: Subacute
Description: Stent/Scaffold Thrombosis (per ARC): Stent/Scaffold Thrombosis should be reported as a cumulative value over time and at various individual time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Subacute stent thrombosis : >24 hours to 30 days after stent implantation
Time Frame: >24 hours to 30 days post stent implantation
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 0

3. Primary Outcome: Number of Participants With Stent Thrombosis: Late
Description: Stent/Scaffold Thrombosis (per ARC): Stent/Scaffold Thrombosis should be reported as a cumulative value over time and at various individual time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Late stent thrombosis : >30 days to 1 year after stent implantation
Time Frame: 30 days to 1 year post stent implantation
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 1

4. Secondary Outcome: Number of Participants With Stent Thrombosis: Very Late
Description: Stent/Scaffold Thrombosis (per ARC): Stent/Scaffold Thrombosis should be reported as a cumulative value over time and at various individual time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Very late stent thrombosis : >1 year after stent implantation.
Time Frame: >1 year post stent implantation
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 0

5. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: The value calculated as 100 * (1- minimum lumen diameter/reference vessel diameter) (MLD/RVD) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Pre-procedure
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions QCA
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Target lesions QCA) | 378
Percent Diameter stenosis | 73.62 (16.20)

6. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: as for outcome 5
Time Frame: post procedure (on day 0)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions QCA
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Target lesions QCA) | 378
Percent Diameter stenosis | 26.03 (12.94)

7. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: as for outcome 5
Time Frame: 8 months
Population: The number of participants analyzed includes subjects who received angiographic follow-up at 8 months.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 226
Number analyzed (Target lesions) | 239
Percent Diameter stenosis | 28.31 (17.02)

8. Secondary Outcome: Success Rate: Percentage of Devices With Implant Success
Description: The stent lengths used were 8 mm, 12 mm, and 15 mm,18 mm, 23 mm, and 28 mm and the stent diameter was 2.25mm.
  Successful delivery and deployment of the first study scaffold/stent the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 50% by quantitative coronary angiography (QCA).
Time Frame: < or = 1 day
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: XIENCE PRIME SV stents
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (XIENCE PRIME SV stents) | 335
percentage of devices | 100 [99.1 to 100]

9. Secondary Outcome: Success Rate: Percentage of Lesions With Procedural Success
Description: Achievement of final in-scaffold/stent residual stenosis of less than 50% by QCA with successful delivery and deployment of at least one study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel MI or repeat TLR during the hospital stay (less than or equal to 7 days).
Time Frame: < or = 1 day
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Lesions) | 326
Percentage of lesions | 100 [99.1 to 100]

10. Secondary Outcome: Success Rate: XIENCE PRIME Implant Success by Patient
Description: The stent lengths used were 8 mm, 12 mm, and 15 mm,18 mm, 23 mm, and 28 mm and the stent diameter was 2.25 mm.
  Implant success is assessed as per physicians decision, but means that the stent could be implanted at the intended location.
Time Frame: < or = 1 day
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
participants | 100 [99.0 to 100.0]

11. Secondary Outcome: Number of Death
Description: Death includes cardiac death, non-cardiac death and non-coronary death.
Time Frame: 0 to 8 months
Population: Intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

12. Secondary Outcome: Number of Death
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  • Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  • Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  • Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: 0 to 1 year
Population: Intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 7

13. Secondary Outcome: Number of Death
Description: as for outcome 12
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 11

14. Secondary Outcome: Number of Death
Description: as for outcome 12
Time Frame: 0-3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 20

15. Secondary Outcome: Number of Death
Description: as for outcome 12
Time Frame: 0-4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 25

16. Secondary Outcome: Number of Death
Description: as for outcome 12
Time Frame: 0-５ years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 30

17. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 2

18. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 17
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 2

19. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 17
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 3

20. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 17
Time Frame: 0-3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

21. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 17
Time Frame: 0-4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

22. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 17
Time Frame: 0-5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 5

23. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: Target lesion revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. Target lesion revascularization (TLR) includes ischemia driven TLR and non-ischemia driven TLR
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 9

24. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: as for outcome 23
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 16

25. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: as for outcome 23
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 22

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: as for outcome 23
Time Frame: 0-3 years
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 25

27. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: as for outcome 23
Time Frame: 0-4 years
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 26

28. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: as for outcome 23
Time Frame: 0-5 years
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 27

29. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: Target vessel revascularization (TLR or TVR, non-TLR) includes ischemia driven TVR (TLR or TVR, non-TLR) or non-ischemia driven TVR (TLR or TVR, non-TLR)
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 21

30. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: as for outcome 29
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 34

31. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: The number of patient with Ischemia-driven Target vessel revascularization (TLR or TVR, non-TLR)
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 42

32. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: as for outcome 29
Time Frame: 0-3 years
Population: ITT popuation
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 45

33. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: as for outcome 29
Time Frame: 0-4 years
Population: ITT popuation
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 47

34. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR, Non-TLR)
Description: as for outcome 29
Time Frame: 0-5 years
Population: ITT popuation
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 51

35. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 16

36. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 32

37. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 42

38. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 45

39. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 55

40. Secondary Outcome: Number of Participants With Non-target Vessel Revascularization (Non-TVR)
Description: Non Target Vessel Revascularization (Non-TVR) is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 58

41. Secondary Outcome: Number of Participants With All Revascularization
Description: Revascularization:
  * Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  * Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  * Non Target Lesion Revascularization (Non-TLR) is any revascularization in the target vessel for a lesion other than the target lesion.
  * Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 34

42. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 41
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 59

43. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 41
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 73

44. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 41
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 78

45. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 41
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 85

46. Secondary Outcome: Number of Participants With All Revascularization
Description: as for outcome 41
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 88

47. Secondary Outcome: Number of Participants With Hemorrhage
Description: Bleeding complications will be defined according to the GUSTO (Global Use of Strategies to Open Occluded Coronary Arteries) classification of severe, moderate, and mild bleeding events.
  Severe or life-threatening:
  Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention
  Moderate:
  Bleeding that requires blood transfusion but does not result in hemodynamic compromise
  Mild:
  Bleeding that does not meet criteria for either moderate or severe bleeding
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 0

48. Secondary Outcome: Number of Participants With Hemorrhage
Description: as for outcome 47
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 1

49. Secondary Outcome: Number of Participants With Hemorrhage
Description: as for outcome 47
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 2

50. Secondary Outcome: Number of Participants With Hemorrhage
Description: Bleeding complications will be defined according to the GUSTO (Global Use of Strategies to Open Occluded Coronary Arteries) classification of severe, moderate, and mild bleeding events.
  Severe or life-threatening: Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention; Moderate: Bleeding that requires blood transfusion but does not result in hemodynamic compromise; Mild: Bleeding that does not meet criteria for either moderate or severe bleeding.
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

51. Secondary Outcome: Number of Participants With Hemorrhage
Description: as for outcome 50
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

52. Secondary Outcome: Number of Participants With Hemorrhage
Description: as for outcome 50
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

53. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 8

54. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 53
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 11

55. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 53
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 16

56. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 53
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 21

57. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 53
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 21

58. Secondary Outcome: Number of Participants With Target Lesion Failure
Description: as for outcome 53
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 25

59. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 38

60. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 66

61. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 84

62. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 96

63. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 106

64. Secondary Outcome: Number of Participants With All Death/All MI/All Revascularization
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 111

65. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: Target vessel failure includes cardiac death, MI, ischemia driven TLR, ischemia driven TVR, non TLR and ischemia driven TVR (TLR or TVR, nonTLR).
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 16

66. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: Target vessel failure includes cardiac death, MI and ischemia driven TLR; ischemia driven TVR, non TLR; ischemia driven TVR (TLR or TVR, nonTLR).
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 22

67. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: as for outcome 66
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 30

68. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: as for outcome 66
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 35

69. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: as for outcome 66
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 39

70. Secondary Outcome: Number of Participants With Target Vessel Failure
Description: as for outcome 66
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 45

71. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and Clinically indicated target lesion revascularization (CI-TLR).
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 9

72. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: as for outcome 71
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 12

73. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: as for outcome 71
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 18

74. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: as for outcome 71
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 23

75. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: as for outcome 71
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 23

76. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: as for outcome 71
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 28

77. Secondary Outcome: Number of Participants With Death or MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 6

78. Secondary Outcome: Number of Participants With Death or MI
Description: as for outcome 77
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 9

79. Secondary Outcome: Number of Participants With Death or MI
Description: All deaths includes Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) Q wave MI Development of new, pathological Q wave on the ECG. Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 14

80. Secondary Outcome: Number of Participants With Death or MI
Description: as for outcome 79
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 22

81. Secondary Outcome: Number of Participants With Death or MI
Description: as for outcome 79
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 27

82. Secondary Outcome: Number of Participants With Death or MI
Description: as for outcome 79
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 33

83. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 5

84. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: as for outcome 83
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 5

85. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: as for outcome 83
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 6

86. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: as for outcome 83
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 8

87. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: as for outcome 83
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 8

88. Secondary Outcome: Number of Participants With Cardiac Death or MI
Description: as for outcome 83
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 12

89. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
Time Frame: 0 to 8 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

90. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel-MI
Description: as for outcome 89
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 5

91. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI
Description: as for outcome 89
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 4

92. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI
Description: as for outcome 89
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 6

93. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI
Description: as for outcome 89
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 6

94. Secondary Outcome: Number of Participants With Cardiac Death or Target Vessel MI
Description: as for outcome 89
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Participants | 9

95. Secondary Outcome: Acute Gain: In-stent,In-segment
Description: The acute gain was defined as the difference between post- and preprocedural minimal lumen diameter (MLD).
Time Frame: Pre procedure to post procedure (on day 0)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Target lesions) | 378
Millimeter
  Stent | 1.56 (0.46)
  Segment | 1.16 (0.48)

96. Secondary Outcome: Late Loss(LL): In-stent,In-segment,Proximal, and Distal
Description: Proximal and distal late loss was calculated by [post-procedure minimum lumen diameter (MLD)] - [MLD at 8 months].
Time Frame: 8 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Target lesions) | 378
Millimeter
  Stent | 0.23 (0.40)
  Proximal | 0.13 (0.32)
  Distal | -0.03 (0.35)
  Segment | 0.09 (0.52)

97. Secondary Outcome: Net Gain: In-stent, In-segment
Description: Difference between acute gain and late loss.
Time Frame: Post-Procedure (on day 0)
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
Number analyzed (Participants) | 312
Number analyzed (Target lesions) | 378
Millimeter
  Stent | 1.31 (0.48)
  Segment | 1.08 (0.52)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | XIENCE PRIME SV Everolimus Eluting Coronary Stent
All-Cause Mortality (participants affected / at risk) | 39/312
Serious Adverse Events (participants affected / at risk) | 165/312
Other Adverse Events (participants affected / at risk) | 0/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE PRIME SV Everolimus Eluting Coronary Stent (N=312)
Anemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 30
Angina unstable (Cardiac disorders) | 10
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery dissection (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 80
Heart failures (Cardiac disorders) | 21
Intracardiac thrombus (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Sick sinus syndrome (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 2
Meniere's disease (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Diverticulitis intestinal hemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3
Inguinal hernia (Gastrointestinal disorders) | 1
Ischemic colitis (Gastrointestinal disorders) | 1
Lower digestive tract haemorrhage (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Death (General disorders) | 8
Cholangitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Bacterial Pneumonia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 9
Anemia postoperative (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 25
Femoral fracture (Injury, poisoning and procedural complications) | 2
Ligament injury (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Cardiac enzymes increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Foot Deformation (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral hemorrhage (Nervous system disorders) | 4
Cerebral infarction (Nervous system disorders) | 10
Syncope (Nervous system disorders) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Coronary revascularisation (Surgical and medical procedures) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 20
Peripheral artery stenosis (Vascular disorders) | 2
Peripheral artery thrombosis (Vascular disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Device related thrombosis (General disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Nephrosis (Renal and urinary disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Pyrexia (General disorders) | 1
Exercise test abnormal (Investigations) | 1
Injury (Injury, poisoning and procedural complications) | 1
Thrombophlebitis (Vascular disorders) | 1
Aortic regurgitation (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Complete AV block (Cardiac disorders) | 1
Prostatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ureter cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Type II diabetes mellitus (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Inner ear disorder (Ear and labyrinth disorders) | 1
Metastatic prostatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoidosis (Immune system disorders) | 2
Ischiadic nerve neuropathy (Nervous system disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Large intestine hemorrhage (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2013-03-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02513719/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT02513719/SAP_001.pdf